CLINICAL TRIAL: NCT05627726
Title: Effectiveness and Cost-effectiveness of PelviSense, a Novel Biofeedback Device With Wearable Sensors for Stress Urinary Incontinence in Women: a Randomised Controlled Trial Alongside Economic Evaluation
Brief Title: Effectiveness and Cost-effectiveness of PelviSense, a Novel Biofeedback Device for Stress Urinary Incontinence in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Priya Kannan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HMRF PolyU
Record Dates: First submitted 2022-11-13; First posted 2022-11-28 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PelviSense-assisted pelvic floor muscle training group (Experimental): Women allocated to the PelviSense-assisted pelvic floor muscle training (PFMT) group will perform PFMT to contract their urethras while the wearable sensors are positioned close to the vagina (to measure pubococcygeus muscle activation). Exercises will be performed in antigravity (supine or side-lying) positions and will progress to against-gravity positions (sitting/ standing).
  Interventions: Device: PelviSense-assisted pelvic floor muscle training group
- Pelvic floor muscle training (PFMT) alone group (Active Comparator): Pelvic floor muscle training (PFMT) alone group: Women allocated to the PFMT alone group will perform unassisted PFMT. Exercise parameters, technique, and progression will be similar to those for the PelviSense-assisted PFMT group, but exercises will be performed without the PelviSense.
  Interventions: Other: Active comparator

INTERVENTIONS:
Device: PelviSense-assisted pelvic floor muscle training group — The PelviSense consists of a high-precision, oval-shaped, wearable EMG sensor that displays electrical activity measured in PFMs on the user's mobile device. The reusable, wearable EMG sensor is non-invasive and can be attached to the user's perineal region. The mobile app provides real-time muscular feedback, displayed as EMG waveforms in microvolts. The mobile app can store data for up to 7 days, allowing participants to monitor their progress over the last 7 days in a graphical format.
  Other Names: Non-invasive novel biofeedback
  Arms: PelviSense-assisted pelvic floor muscle training group
Other: Active comparator — Pelvic floor muscle training (PFMT) alone group: Women allocated to the PFMT alone group will perform unassisted PFMT. Exercise parameters, technique, and progression will be similar to those for the PelviSense-assisted PFMT group, but exercises will be performed without the PelviSense.
  Other Names: Pelvic floor muscle training (PFMT) alone group
  Arms: Pelvic floor muscle training (PFMT) alone group

SUMMARY:
Aims: (1) Investigate the efficacy of PelviSense-assisted PFMT compared with PFMT alone for improving SUI symptom severity in women; (2) Compare the cost-effectiveness of the PelviSense device against PFMT alone for treating SUI in women; (3) Explore the views of women regarding the use of the PelviSense device as an adjunct to PFMT and the impacts of the PelviSense device on their lives and well-being.

Design and subjects: A sequential, embedded, experimental mixed-methods design, including a randomised controlled trial (RCT) and semi-structured focus groups, will be conducted alongside an economic evaluation. The proposed study will include 142 women with SUI or stress-predominant mixed urinary incontinence.

Interventions: Women will be randomly allocated to one of two groups (PelviSense or PFMT alone [control]). The PelviSense group will perform PFMT with assistance from the PelviSense device, and the control group will perform PFMT without biofeedback (i.e., PFMT alone).

Outcome measures: International Consultation on Incontinence Questionnaire-Short Form, one-hour pad test, Modified Oxford Scale, EQ-5D-5L, and electronic cost diary.

Data analysis and expected results: Statistical analysis will be conducted using analysis of covariance. The PelviSense group is expected to report significant improvements in primary and secondary outcomes compared with the PFMT alone group. The PelviSense group will yield cost savings and result in lower health care utility compared with the PFMT alone group.

DETAILED DESCRIPTION:
Background Pelvic floor muscle (PFM) training (PFMT) is a common conservative first-line treatment for SUI in women. However, the success of PFMT alone, without adjunctive therapies, has been hampered by the lack of training adherence among patients, who report the inability to contract the correct PFMs and limited motivation to perform PFMT exercises. Therefore, PFMT is often combined with adjunctive therapies, such as electromyography (EMG) biofeedback via an intravaginal probe (referred to as conventional biofeedback), transvaginal electrical stimulation (TVES), or weighted vaginal cones. However, PFMT adjunctive therapies that involve intravaginal probes/ cones are not preferred by women because they are invasive, and the vaginal insertion of probes/ cones can cause pain and discomfort. In addition, older women with atrophic vaginas have difficulty retaining probe/cones within the vaginal canal due to weak PFM tone.

To meet the existing need for a non-invasive PFMT adjunctive therapy, the research team developed the PelviSense. The PelviSense is an innovative, non-invasive biofeedback device with wearable EMG sensors, designed to assist individuals in isolating and strengthening PFMs by helping them distinguish correct PFM contractions (lifting or squeezing the muscles) from incorrect attempts (bearing down). A mixed-methods study, including a full-scale RCT and semi-structured focus groups, alongside an economic evaluation, will be conducted to evaluate both the effectiveness and cost-effectiveness of the newly developed PelviSense device for the treatment of SUI in women.

Aims:

Aim 1: Investigate the efficacy of PelviSense-assisted PFMT compared with PFMT alone for improving SUI symptom severity in women.

Aim 2: Compare the cost-effectiveness of the PelviSense device against PFMT alone for treating SUI in women.

Aim 3: Explore the views of women regarding the use of the PelviSense device as an adjunct to PFMT and the impacts of the PelviSense device on their lives and well-being.

Methods Recruitment: Women with SUI who attend the outpatient Obstetrics and Gynecology Department of Kwong Wah Hospital (KWH) will be recruited for the study. In addition, potential participants will be recruited using a non-probability convenience sampling technique through public, KWH, elderly care centers, and HK Polytechnic University (PolyU) campus advertising. Advertising will consist of study flyers posted at KWH, around the university campus, in waiting rooms of university health services and physiotherapy clinics, in community churches, and in university-owned amenities, including sports centres and gyms.

Randomisation and blinding: Computer-generated randomisation will be utilised to ensure that both study groups are assigned an equal number of participants at a 1:1 ratio. Sequentially numbered, sealed, opaque envelopes of similar size and shape will be utilised to conceal group allocation and avoid selection bias. Due to the nature of the intervention, it is not possible to blind the therapists or participants to the allocation of treatment; therefore, only the outcome assessor will be blinded. To minimise detection bias, the outcome assessors will not participate in the treatment, and all study outcomes will be assessed in a separate room without any knowledge of participant allocation. Statistical analysis will be performed in a blinded manner, with each group assigned a code (group A and group B). The group identities will be revealed after all analyses are completed.

Procedure and baseline assessment: Potentially eligible women who contact research personnel will be invited to attend an in-person screening session. On this first day of contact, all women will undergo BMI measurement; complete the screening questionnaire, MMSE, and 1-h pad test to confirm eligibility; and provide written informed consent. Baseline assessments of study outcomes will be performed, and eligible and consenting participants will be randomised to intervention groups.

Outcome measures Outcomes assessments will be completed at baseline (time point 1 [T1]), 1-month (T2) and 6-months (T3).

Intervention. The interventions will be provided for 6 months, beginning with a 1-month supervised training period at KWH and PolyU. Following supervised training, women will be instructed to perform unsupervised home exercises for 5 months. Unsupervised home exercises will consist of at least eight contractions, performed 3 times per day, for 5 days of each week, with or without the biofeedback device according to group assignment. Each contraction will last for 10 seconds, followed by relaxation for 10 seconds. The PFMT exercise parameters are based on the National Institute for Health and Care Excellence PFMT guidelines for UI.

Qualitative study (semi-structured focus groups). A computer-generated randomization schedule will be utilized to identify 20 participants (from the 71 participants included in the PelviSense-assisted PFMT group) to participate in the focus groups. Each focus group will last for 45-60 minutes. Focus groups will continue to be conducted until data saturation occurs. Focus groups will be scheduled for 8-months post-randomisation. A semi-structured focus group approach will be used, during which discussion will be guided by but not limited to a set of pre-determined, open-ended questions.

Data processing and analysis: Statistical analysis will be performed on an intention-to-treat basis using the Statistical Package for the Social Sciences (v.25; Armonk, NY).

Treatment effects for both primary and secondary outcomes between T1, T2, and T3 and across the intervention groups will be evaluated using a two-way analysis of covariance (ANCOVA) with age as the covariate. T1 and T2 will be compared to establish immediate treatment effects, and T1 and T3 will be compared to evaluate the retention of treatment effects. For significant group by time interaction effects, post-hoc analysis using Bonferroni correction will be performed.

The unadjusted mean total and disaggregated costs and differences in costs between the PelviSense and PFMT alone groups will be calculated. Seemingly unrelated regression (SUR) analyses will be used to estimate total cost differences (ΔC) and effect differences (ΔE).

The EQ-5D-5L responses will be converted into utility scores to estimate the gain or loss of quality-adjusted life-years (QUALYs). The incremental cost-effectiveness ratio (ICER) will be calculated using the formula ICER = ΔC / ΔE. Uncertainty surrounding ICERs and 95% confidence intervals for cost differences will be estimated using bias-corrected and accelerated bootstrapping with 5,000 replications.

Qualitative data from the focus groups will be analysed using the six phases of thematic analysis recommended by Braun and Clarke. The identified themes will then be defined and named according to their contents. The final set of themes will be confirmed as coherent and comprehensive by review of the team.

ELIGIBILITY:
Inclusion Criteria:

* non-pregnant women with stress urinary incontinence (SUI),
* aged 35 to 65 years,
* women who experience mild to moderate SUI, as indicated by a pad weight gain of 1-50 g during the 1-hour pad test with stress test,
* women with a score ≥24 on the Mini-Mental State Examination.

Exclusion Criteria:

* women <6 months postpartum,
* women with severe pelvic organ prolapse,
* women with complicated SUI due to pelvic region radiation,
* women with a body mass index (BMI) ≥30,
* women with severe psychological problems impairing study participation,
* women with mixed urinary incontinence (MUI) or urge urinary incontinence (UUI)

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
Stress urinary incontinence (SUI) symptom severity | Baseline (0 month)
  (ICIQ-SF) will be used to measure SUI symptom severity.
Stress urinary incontinence (SUI) symptom severity | 1-month
  The disease-specific International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) will be used to measure SUI symptom severity.
Stress urinary incontinence (SUI) symptom severity | 6 months
  (ICIQ-SF) will be used to measure SUI symptom severity.

SECONDARY OUTCOMES:
The severity of urine leakage | Baseline (0 month)
  The one-hour (1-h) pad test will be used to quantify the severity of urine leakage.
The severity of urine leakage | 1-month
  The one-hour (1-h) pad test will be used to quantify the severity of urine leakage.
The severity of urine leakage | 6 months
  The one-hour (1-h) pad test will be used to quantify the severity of urine leakage.
Pelvic floor muscle strength | Baseline (0 month)
  The valid and reliable Modified Oxford Scale (MOS) will be used to grade PFM.
Pelvic floor muscle strength | 1-month
  The valid and reliable Modified Oxford Scale (MOS) will be used to grade PFM.
Pelvic floor muscle strength | 6 months
  The valid and reliable Modified Oxford Scale (MOS) will be used to grade PFM.
Economic evaluation | 1-month
  The cost for private health services will be estimated using self-reported data collected from the Client Service Receipt Inventory (CSRI) form.
Economic evaluation | 6-months
  The cost for private health services will be estimated using self-reported data collected from the Client Service Receipt Inventory (CSRI) form.
Quality-adjusted life-years (QUALYs) | 1-month
  The EQ-5D-5L will be used to evaluate health-related quality of life (QoL) for the PelviSense and PFMT alone groups.
Quality-adjusted life-years (QUALYs) | 6 months
  The EQ-5D-5L will be used to evaluate health-related quality of life (QoL) for the PelviSense and PFMT alone groups.

CONTACTS AND LOCATIONS:
Overall Officials: PRIYA KANNAN, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong
  - Kwong Wah Hospital, Kowloon

IPD SHARING:
Plan to Share IPD: No
Data will be made available on request